CLINICAL TRIAL: NCT02893319
Title: Role of Infant Feeding, Childhood Food Habits and Early Childhood Adiposity (RIF)
Brief Title: Maternal and Infant Growth Study
Acronym: RIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leann Birch (Other)
Responsible Party: Sponsor-Investigator, Leann Birch, William P. Flatt Professor, University of Georgia
Organization: University of Georgia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013102510
Record Dates: First submitted 2016-08-24; First posted 2016-09-08 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Maternal Behavior; Body Weight; Infant Behavior
Keywords: Infant Feeding; Infant Growth
MeSH Terms: conditions — Body Weight; Infant Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breastfeeding (No Intervention): control group
- 5 oz bottle (Active Comparator): Subject will feed infant with 5oz medela bottle
  Interventions: Behavioral: Feeding and growth differences, 5oz vs 8oz bottle
- 8 oz bottle (Active Comparator): Subject will feed infant with 8oz medela bottle
  Interventions: Behavioral: Feeding and growth differences, 5oz vs 8oz bottle

INTERVENTIONS:
Behavioral: Feeding and growth differences, 5oz vs 8oz bottle — Group A: 5oz bottle Group B: 8oz bottle
  Arms: 5 oz bottle; 8 oz bottle

SUMMARY:
Rapid growth early in infancy is a risk factor for obesity and cardiovascular disease later in the lifespan. Evidence is limited, but both pre- and postnatal factors are associated with early rapid growth, and include high maternal BMI prior to pregnancy and excessive gestational weight gain. This research focuses on aspects of early feeding as potentially modifiable factor affecting early infant weight gain. Formula feeding mothers are randomized to receive either 5 oz of 8 oz bottles to use in feeding their infants from 2- to 16 weeks postpartum. In addition, a reference group of exclusively breastfeeding mother-infant dyads are also included. The hypothesis is that differences in feeding practices will be associated with differences in growth and that infants randomized to be fed from smaller bottles will grow more slowly that those randomized to larger bottles. Growth patterns of formula fed infants will also be compared to those of exclusively breastfed infants.

DETAILED DESCRIPTION:
Mothers complete feeding logs, questionnaires on health history, demographics, feeding attitudes and practices. Infant growth and body composition are measured via PEA POD, and maternal anthropometrics and body composition are measured in BOD POD the laboratory at 2, 8, and 16 weeks postpartum. Primary outcome is change in weight-for-age z-scores.

ELIGIBILITY:
Inclusion Criteria:

* pregnant or newborn aged 28 days or younger

Exclusion Criteria:

* gestational diabetes, hypertension, pregnancy/delivery complications, premature birth, low birth weight

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in Infant Weight-for-Age Z-score over time by group | 2, 8 and 16 weeks of age
  Infant weight (kg) (PEA POD scale) will be measured at each of three time points (2, 8, 16 weeks of age). Weight-for-Age Z-score (WAZ) will be calculated based on World Health Organization Global Database on Child Growth, means will be calculated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Leann L Birch, PhD, Principal Investigator — The University of Georgia

IPD SHARING:
Plan to Share IPD: No
All data is de-identified.